CLINICAL TRIAL: NCT06959576
Title: Microbial and Laboratory Study of 3D-Printed Reinforced Acrylic Denture
Brief Title: Trueness and Dimensional Deviation of 3D Printed Nanocomposite Maxillary Denture Base Resin (In Vivo Study)
Acronym: dimensions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Eman Mohamed Teama, Principal investigator, Tanta University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: RP 2#23 1
Record Dates: First submitted 2025-04-16; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Denture Hyperplasia
Keywords: 3Dprinted denture base; nanoparticles; trueness; dimensional deviation
MeSH Terms: interventions — Nanoparticles

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nanoparticles (Other): Nanoparticles improve the quality of 3D-printed denture base resin
  Interventions: Other: nanoparticles

INTERVENTIONS:
Other: nanoparticles — Nanoparticles improve the dimensional stability of 3D printed denture base resin, so preventing instability of the denture over time
  Other Names: ZrO2; TiO2

SUMMARY:
Purpose: To evaluate the effect of adding nano ZrO2 and nano TiO2 nanoparticles on trueness and dimensional deviation of maxillary 3D printed denture base resin on completely edentulous patients.

Materials and Methods: This study was carried out on 24 completely edentulous patients. The patients were divided randomly into three equal groups; Group I: Patients received 3D printed maxillary complete denture without additives, Group II: Patients received 3D printed maxillary complete denture reinforced by Nano ZrO2 (0.4%) by Wt and Group III: Patients received 3D printed maxillary complete denture reinforced by Nano TiO2 (0.4%) by Wt. Trueness was evaluated by scanning the denture using an extraoral scanner after the printing process, before insertion. Dimensional deviation was evaluated by scanning the denture using an extraoral scanner at the time of insertion and after 6 months, 12 months, and 18 months. The trueness and dimensional deviation values were analyzed using repeated measure ANOVA, followed by multiple comparison Turkey test.

DETAILED DESCRIPTION:
* Primary and final impressions of the maxillary and mandibular arches were taken for each patient following basic prosthetic principles.
* Maxillary and mandibular record blocks were made on the master casts and adjusted in the oral cavity of the patients in a normal manner to ensure an acceptable vertical dimension at occlusion and a freeway space of 2-4 mm. The centric relationship was recorded via the static method.
* An extra-oral scanner was used for scanning master casts (upper and lower), then occlusion blocks on the master cast were scanned after spraying with the scanner spray.
* Master casts and jaw relation records. Standard tessellation language (STL) files were sent to the software platform (Exocad). The software enabled virtually simultaneous mounting and alignment.
* Virtual design of the upper and lower bases and virtual setting of the upper and lower teeth were performed.
* The virtual denture STL file was exported to the LCD printer, which prints the denture base and teeth (trial base) as one unit.
* The try-in step was performed via the trial denture base to check for occlusion, esthetics, and denture border extension.

If any modification was performed on teeth using articulating paper or in the denture base using pressure-indicating paste, the trial denture bases were scanned by an extraoral scanner. The STL file was then sent again to the software for correction of the design, and then sent to the 3D printer software.

* Before printing, each file was checked for support adequacy, the printing orientation was 45 degrees, the thickness of the printed layer was 50 microns, and the printing time was 4 hours and 7 seconds for each denture15
* The denture base and the teeth were printed separately via a 3D printer.16
* For Group Ι, Pink denture base resin was used without nanoparticles for printing the denture bases. However, for Group II, Pink denture base resin reinforced by nanoparticles (ZrO2) (0.4%) by weight was used for printing the denture bases.
* Additionally, for Group III, pink denture base resin reinforced with nanoparticles (TiO2) (0.4%) by weight was used for printing the denture bases.
* For printing the teeth, white tooth resin was used for all groups.
* To remove any residual monomers after printing, the denture bases and teeth were placed in isopropyl alcohol for five minutes.
* Finally, resin was used to attach teeth to recessed pockets in the denture bases, after which the dentures were placed in the postcuring unit.
* Eventually, the dentures were finished, and the teeth were coated with resin glaze to protect and polish areas of posterior pits and fissures and interproximal surfaces from staining or discoloration.
* The dentures were inserted into the patient's mouth and checked for any necessary adjustments, and every patient was given the same post-insertion instructions for home care and follow-up evaluation, and a regular oral and denture hygiene protocol.

ELIGIBILITY:
Inclusion Criteria:

All patients participating in this study were selected according to the following criteria:

* Completely edentulous patients with good local and systemic health.
* With an age range of 50 to 70 years old.
* Have adequate interarch space and class Ⅰ angle classification.
* Have good neuromuscular control. Patient exclusion criteria
* Any disease that may affect denture construction
* Oral parafunctional habits.
* Temporomandibular disorders

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Trueness of 3D printing | After printing 0 days
  Scanning of the maxillary denture bases was done using the extraoral scanner.
  * Each denture was sprayed by scanning spray and was placed on the scanning table. The STL files were saved for evaluation. The STL file of each 3D printed denture base was compared with the STL file of the original design.
  * A 3D analysis software (Medit link) and root mean square (RMS) calculation method were used to evaluate the deviations of the maxillary denture bases when compared with the original STL file. Original STL file and test-STL files were imported into the software, and the original STL was selected as the reference.
  * Test-STL was superimposed over the original STL by using the comparison tool of the software, which allows simultaneous selection of 3 points on both files.
  * Software automatically calculated overall RMS values; thus, no additional formula was used. Color-difference maps were generated to calculate the RMS values.
Dimensional deviation of maxillary 3D printed denture base resin | 18 months
  Evaluation was carried out during the time of insertion, after 6,12and 18 months.
  * Maxillary dentures were placed over an acrylic index and fixed to the rotary table of the desktop scanner by using sticky wax.
  * The scanning procedure was done from various angles to obtain both the fitting and polished surface of the denture. The produced STL file from the first scan was saved as a baseline or master file for the subsequent measurements.
  * At 6,12, and 18 months, the denture was scanned again, and at each time the resultant STL file was superimposed on the master file to obtain color maps of dimensional deviation using Medit Link software.
  * Eight areas of interest for the accuracy evaluation of dentures were defined at the intaglio surface: right and left edentulous crests, right and left buccal flanges, central palate, postdam, and right and left tuberosity, with average points selected from each area.

CONTACTS AND LOCATIONS:
Overall Officials: Houda Amin Rashad, prof, Study Director — Tanta University; Eman Mohamed Shakal, prof, Study Director — Tanta University
Locations (1):
- Faculty of dentistry Tanta university Egypt, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Following the research ethics committee of the faculty of dentistry Tanta university